CLINICAL TRIAL: NCT00909961
Title: A One Year, Local, Open Label, Multicentre Trial Evaluating the Effects of Zoledronic Acid 5 mg Infusion on BMD and Biochemical Markers of Bone in PMO Pts Between the Ages of 50 and 65 Years
Brief Title: A Trial Evaluating the Effects of Zoledronic Acid 5 mg Infusion on Bone Mineral Density (BMD) in Postmenopausal Osteoporosis (PMO) Patients Between the Ages of 50 and 65 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446HTR04
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Osteoporosis; Bone Mineral Density; Biomarkers
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Zoledronic Acid

ARMS (1):
- Zoledronic acid (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
This study will evaluate the effects of zoledronic acid 5 mg infusion on BMD and biochemical markers of bone in post-menopausal osteoporotic patients aged between 50-65.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal osteoporosis
* Patients who has a low bone mineral density at hip or vertebral
* Patients who has an osteoporotic fracture at hip or vertebra

Exclusion Criteria:

* Hypersensitivity either to the active substance or to any of the excipients or to any biphosphonates.
* Known metabolic bone disease excluding osteoporosis.
* Serious systemic disorder treated with drugs interfering with bone metabolism.
* Significant liver or renal failure
* Pathologic fracture in the examined body area or elsewhere.
* Previous anti-osteoporotic treatment within 12 months or less prior to the recruitment.
* Patients with hypocalcaemia

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12-16 (Actual)

PRIMARY OUTCOMES:
Efficacy - BMD | 1 year

SECONDARY OUTCOMES:
Efficacy - Biochemical markers | 6 months
Safety - Rate of adverse events and serious adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Turkey (Türkiye) (6):
  - Novartis Investigational site, Ankara
  - Novartis Investigative site, Antalya
  - Novartis Investigational site, Istanbul
  - Novartis Investigative site, Izmir
  - Novartis Investigative site, Kayseri
  - Novartis Investigative site, Konya